CLINICAL TRIAL: NCT03522376
Title: Diaphragm and Sternocleidomastoid Muscle Activation Patterns During Different Loaded Inspiratory Muscle Performance in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Inspiratory Muscle Activation Patterns in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201802054RINB
Record Dates: First submitted 2018-03-25; First posted 2018-05-11 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2018-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic obstructive pulmonary disease: Subjects with the diagnosis of chronic obstructive pulmonary disease, stable clinically, has no infection or acute exacerbation in the previous four weeks, and can cooperate with the measurements of this study, loaded inspiratory muscle test.
  Interventions: Other: Loaded inspiratory muscle test

INTERVENTIONS:
Other: Loaded inspiratory muscle test — Loaded inspiratory muscle tests will be set at 30% and 50% of maximal inspiratory pressure. The orders of the two loaded test conditions will be conducted in random order with at least 24 hours separation. This is an observational study. Subjects will perform only 15 breaths with each loaded test condition to exam the performance of their inspiratory muscles. Loaded inspiratory muscle test is not for training.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a chronic inflammatory lung disease that causes obstructed airflow from the lung, characterized by chronic cough, dyspnea, and sputum production. Inspiratory muscle weakness has been shown in patients with COPD, and inspiratory muscle training (IMT) is commonly applied to these patients. However, the optimal prescribed intensity of IMT for patients with COPD remains unclear. In healthy adults the accessory muscles would be recruited to assist ventilation with increasing ventilatory demand, but the activation pattern of accessory muscles has not been studied in patients with COPD during loaded condition such as IMT. Therefore, the purpose of this study is to exam diaphragm and sternocleidomastoid muscle activation using surface electromyography during loaded inspiratory muscle tests with intensity of 30% and 50% of maximal inspiratory pressure.

DETAILED DESCRIPTION:
The prevalence of chronic obstructive pulmonary disease (COPD) is 11.7% around the world in 2010, and it is expected to rise over the next 30 years. COPD is a chronic inflammatory lung disease that causes obstructed airflow from the lung, characterized by chronic cough, dyspnea, and sputum production. Studies have found evidences of inspiratory muscle weakness in patients with COPD which include a reduction in maximal inspiratory pressure (PImax), a shift toward oxidative type I fibers and atrophy in all types of fibers in diaphragm muscle. The shift of diaphragm muscle fiber toward oxidative type I fibers might result from endurance training-like effect that served to counteract the negative effects of elevated oxidative stress and systemic inflammation in patients with COPD.

Inspiratory muscle training (IMT) is commonly applied to patients with COPD during pulmonary rehabilitation, but its clinical benefits remain inconclusive. Some studies showed that IMT improves breathing pattern, dyspnea and the strength and endurance of diaphragm, while others showed that IMT could not improve inspiratory muscle strength and functional exercise capacity either applied alone or in addition to pulmonary rehabilitation in patients with COPD. Evidence from animal study showed that overloading the diaphragm during resistive breathing might induce acute diaphragm injury. Increases oxidative stress and systemic inflammation, and exacerbating the apoptosis of the diaphragm fibers may also occur during IMT in patients with COPD, which leads to the progression of diaphragm muscle fibers atrophy. In human studies, the intensity used for IMT ranged from 10% to 70% of PImax, and the training effect showed no clear dose-response pattern. The optimal intensity that would induce positive physiological effect without eliciting overloading injury remains unclear. In healthy adults, the accessory muscles, such as sternocleidomastoid (SCM), scalenes, and intercostals muscle, would be recruited to assist ventilation with increasing ventilatory demand. Thus the activation of accessory muscles could be an indicator for training overload. However, the activation pattern of accessory muscle has not been studied in patients with COPD during IMT. Whether the commonly prescribed intensity for IMT would lead to excessive activation of diaphragm, and more accessory muscle recruitment in patients with COPD remains to be determined. Therefore, the purpose of this study is to exam diaphragm and SCM muscle activation using surface electromyography during loaded inspiratory muscle tests with 30% and 50% of PImax intensity.

ELIGIBILITY:
Inclusion Criteria:

* age > 20 years old
* has been diagnosis of chronic obstructive pulmonary disease with stable clinical condition with no infection or acute exacerbation in the previous four weeks
* can cooperate with the measurements of this study

Exclusion Criteria:

* any clinical diagnosis that will influence the measurement, including any history of neuromyopathy
* angina, acute myocardial infarction in the previous one month
* pregnancy
* participated in inspiratory muscle training program in the previous three months
* any psychiatric or cognitive disorders, for example: Mini-Mental State Examination (MMSE) < 24, that will disturb the communication and cooperation of the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic obstructive pulmonary disease is a chronic inflammatory lung disease that causes obstructed airflow from the lung, characterized by chronic cough, dyspnea, and sputum production. Recent studies show that other than respiratory symptoms, patients with chronic obstructive pulmonary disease often present with inspiratory muscle weakness.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Diaphragm and Sternocleidomastoid muscle activation | through the completion of the loaded inspiratory muscle test condition; it would take about 3 minutes
  Root mean square values during different conditions
The mean median frequency of diaphragm and sternocleidomastoid muscle | In one minute after the completion of the loaded inspiratory muscle test condition
  The power spectrum is divided into two equal areas of the frequency value by median frequency to exam muscle fatigability

CONTACTS AND LOCATIONS:
Overall Officials: Li-Ying Wang, Phd, Study Chair — National Taiwan University
Locations (1):
- School and Graduate Institute of Physical Therapy of National Taiwan University, Taipei, Zhongzheng Dist, Taiwan